CLINICAL TRIAL: NCT06565117
Title: Efficacy of Dipotassium Glycyrrhizinate Emollients in the Maintenance Treatment of Adult Atopic Dermatitis: A Single-Center Randomized Controlled Study
Brief Title: Efficacy of Dipotassium Glycyrrhizinate Emollients in the Maintenance Treatment of Adult Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2022-KL323-02
Record Dates: First submitted 2024-08-18; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Adult Atopic Dermatitis
Keywords: Adult Atopic Dermatitis; Efficacy of Dipotassium Glycyrrhizinate Emollients
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A:Emollient for systemic application (Experimental): Emollient for systemic application
  Interventions: Drug: White yu green skin lotion
- B:Emollient was applied locally (Experimental): Apply skin lotion in locally affected skin areas or in areas previously affected by AD
  Interventions: Drug: White yu green skin lotion
- C:No moisturizer (No Intervention): No moisturize

INTERVENTIONS:
Drug: White yu green skin lotion — Group A: Systemic emollient was applied twice daily for 8 weeks Group B: Continue applying skin lotion twice daily in locally affected skin areas or in areas previously affected by AD for 8 weeks
  Arms: A:Emollient for systemic application; B:Emollient was applied locally

SUMMARY:
To investigate whether emollients containing dipotassium glycyrrhizinate have a sustained improvement in the clinical severity of mild to moderate atopic dermatitis in adult.

DETAILED DESCRIPTION:
Atopic dermatitis (atopic eczema, AD) is a common skin inflammatory disease, dry skin and itchy skin is a significant symptom of most AD, often accompany patients for life, seriously affecting the physical and mental health and work life of patients. The number of AD patients is increasing worldwide, while the prevalence rate in China has increased more significantly in the past 10 years. It is characterized by persistent skin dryness and a reduced function of the skin as a barrier to the external environment. Encourage the free use of moisturizers (emollients) as a baseline treatment for AD and add anti-inflammatory therapy as needed. Currently, topical corticosteroids are still the first-line treatment options. However, studies have confirmed that patients with AD are cautious about the use of topical corticosteroids. Maintaining the humidity of the skin and restoring the barrier function of the skin is the basis of the treatment of atopic dermatitis. And studies have shown that regular use of emollients can improve skin hydration, restore the skin barrier, reduce the frequency of attacks, and reduce the use of topical corticosteroids. In patients with AD, daily use of moisturizing emollients enhances the response to topical corticosteroid therapy, reduce percutaneous water loss (TEWL), restore the skin barrier and promote hydration, and can prevent or reduce AD attacks by improving the associated skin barrier defects, prolonging the time between AD episodes. The purpose of this study is to see whether emollients have sustained improvement on the clinical severity of adult atopic dermatitis in maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Williams diagnostic criteria
* SCORAD scores < 50 points, classified according to the severity levels of SCORAD scores, where scores of 0-25 are categorized as mild, and scores of 26-50 are categorized as moderate
* No gender limit, age between 18-65 years old.

Exclusion Criteria:

* Acute disease with erosion, exudation, secondary infection
* There are currently other active inflammatory skin diseases
* Antihistamine was used within 2 weeks prior to enrollment
* Patients treated with emollients and receiving topical drugs (such as glucocorticoids and calcineurin inhibitors) within 1 week before enrollment
* Patients have used phototherapy, systemic corticosteroids, immunosuppressants (such as cyclosporine, azathioprine, or immunoglobulin, etc.) within 4 weeks before enrollment
* The systematic withdrawal time of biological agents or JAK inhibitor (dupilumab, omalizumab, et al) was less than 12 weeks
* Malignant tumors, chronic systemic diseases (such as diabetes mellitus, hypothyroidism), or other acute and chronic infections
* Those known to be allergic to the ingredients of emollient or Hydrocortisone cream
* Patients who have attended or are attending other clinical investigators within three months
* Patients judged unsuitable by the investigator to participate in this study.

Ages: 17 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
SCORAD | Before treatment, Treatment for 2 weeks, 4 weeks, and 8 weeks
  Objective severity of the clinical signs of atopic dermatitis
POEM | Before treatment, Treatment for 2 weeks, 4 weeks, and 8 weeks
  Patient-oriented eczema measurement scores
NRS | Before treatment, Treatment for 2 weeks, 4 weeks, and 8 weeks
  Pain digital score
ADCT | Before treatment, Treatment for 2 weeks, 4 weeks, and 8 weeks
  Long-term disease control
DLQI | Before treatment, Treatment for 2 weeks, 4 weeks, and 8 weeks
  Quality of life index in dermatology

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No